CLINICAL TRIAL: NCT04871529
Title: Randomized Phase II Trial of Gemcitabine, Avelumab and Carboplatin vs. No Neoadjuvant Therapy Preceding Surgery for Cisplatin-Ineligible Muscle-Invasive Urothelial Carcinoma: SWOG GAP TRIAL
Brief Title: Testing the Addition of an Anti-Cancer Immunotherapy Drug, Avelumab, to Gemcitabine and Carboplatin Chemotherapy Prior to Surgery in Muscle Invasive Urinary Tract Cancer vs. Surgery Alone in Patients Who Are Not Able to Receive Cisplatin Therapy (SWOG GAP TRIAL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to accrue sufficient patients
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2011; NCI-2021-02265 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Bladder Carcinoma Infiltrating the Muscle of the Bladder Wall; Infiltrating Renal Pelvis and Ureter Urothelial Carcinoma; Stage II Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — avelumab; B7-H1 Antigen; Gemcitabine; Carboplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (avelumab, gemcitabine, carboplatin, surgery) (Experimental): Patients receive avelumab IV over 60 minutes on day 1. Treatment repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up 4 in the absence of disease progression or unacceptable toxicity. Within 4-8 weeks after final systemic therapy, patients undergo standard of care surgery.
  Interventions: Procedure: Therapeutic Conventional Surgery; Drug: Avelumab; Drug: Gemcitabine Hydrochloride; Drug: Carboplatin
- Arm B (surgery) (Experimental): Patients undergo standard of care surgery.
  Interventions: Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: Avelumab — Given IV
  Other Names: 1537032-82-8; Bavencio; Immunoglobulin G1-lambda1; Anti-(Homo sapiens CD274 (Programmed Death Ligand 1, PDL1, pd-l1, B7 Homolog 1, B7H1)); Homo sapiens Monoclonal Antibody; MSB-0010718C; MSB0010718C
  Arms: Arm A (avelumab, gemcitabine, carboplatin, surgery)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: 1-(2-Oxo-4-amino-1,2-dihydropyrimidin-1-yl)-2-deoxy-2,2-difluororibose, hydrochloride; 122111-03-9; 2''Deoxy-2'',2''-Difluorocytidine Hydrochloride; dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
  Arms: Arm A (avelumab, gemcitabine, carboplatin, surgery)
Drug: Carboplatin — Given IV
  Other Names: (SP-4-2)-diammine[1,1-cyclobutanedicarboxylato(2--)-O,O'']platinum; 1,1-cyclobutanedicarboxylic acid platinum complex; 41575-94-4; Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; cis-diammine(1,1-cyclobutanedicarboxylato) platinum(II); Cis-Diammine(cyclobutane-1,1-dicarboxylato)platinum; cis-diammine(cyclobutanedicarboxylato)platinum II; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; platinum; diammine(1,1-cyclobutanedicarboxylato(2-))-, (SP-4-2)
  Arms: Arm A (avelumab, gemcitabine, carboplatin, surgery)

SUMMARY:
This phase II trial studies the effect of avelumab, gemcitabine and carboplatin before surgery compared with surgery alone in treating patients with muscle invasive bladder or upper urinary tract cancer who are not able to receive cisplatin therapy. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as gemcitabine and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving avelumab together with gemcitabine and carboplatin before surgery may work better in lowering the chance of muscle invasive urinary tract cancer growing or spreading, in patients who cannot receive cisplatin therapy compared to surgery alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare pathologic complete response (pCR, pT0N0) with avelumab plus gemcitabine and carboplatin (AGCa) versus (vs.) no neoadjuvant therapy preceding protocol surgery for muscle-invasive bladder cancer or upper tract urothelial carcinoma (MIBC/UTUC) for participants who are ineligible for cisplatin-based chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate toxicities with AGCa, and to compare resectability rates and surgical complications by arm in this population.

II. To compare event-free survival (EFS) with AGCa versus no neoadjuvant therapy in this population.

III. To compare overall survival (OS) with AGCa versus no neoadjuvant therapy preceding surgery in this population.

IV. To compare pathologic complete response (pCR, pT0N0) with avelumab plus gemcitabine and carboplatin (AGCa) vs. no neoadjuvant therapy preceding protocol surgery in the subset of participants who received at least 2 cycles of neoadjuvant therapy in Arm A.

BANKING OBJECTIVE:

I. To bank tumor tissue, blood, and urine for future correlative genomic, transcriptomic, and proteomic studies to discover molecular signatures associated with pCR and resistance.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive avelumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up 4 in the absence of disease progression or unacceptable toxicity. Within 4-8 weeks after final systemic therapy, patients undergo standard of care surgery.

ARM B: Patients undergo standard of care surgery.

After completion of study treatment, patients are followed up every 12 weeks for years 1-2, every 6 months for year 3, then annually in years 4-5.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have one of the following:

  * Histologically documented muscle-invasive bladder carcinoma (MIBC) from transurethral resection of bladder tumor (TURBT) within 56 days prior to registration
  * Histologically confirmed high grade upper tract urothelial carcinoma (UTUC) within 56 days prior to registration, with invasion confirmed by either a mass on cross-sectional imaging or a tumor directly visualized during upper urinary tract endoscopy within 56 days prior to registration
  * Participants diagnosed with mixed urothelial carcinoma and variant histology within 56 days prior to registration may be eligible if the majority (> 50%) of the tumor consists of urothelial carcinoma. Participants with pure non-urothelial variant histologies or any small cell histology are not eligible
* Participants must have clinical stage T2-T4aN0M0 bladder or upper tract cancer confirmed by radiologic staging (computed tomography [CT] scan/magnetic resonance imaging [MRI] abdomen and pelvis, and CT scan/x-ray of the chest) within 56 days prior to registration
* Participants must have a bone scan within 56 days prior to registration if they have bone pain or elevated serum alkaline phosphatase
* Participants must have a bimanual examination under anesthesia within 56 days prior to registration
* Participants must not have received prior systemic chemotherapy, immunotherapy or radiotherapy for the treatment of muscle invasive bladder cancer (MIBC) or upper tract urothelial carcinoma (UTUC). Other prior pelvic radiotherapy is allowed if it does not preclude surgery (radical cystectomy, nephroureterectomy or ureterectomy, based on location of primary tumor). Prior intravesical therapy is allowed
* Participants must not have received immunosuppressive medication within 14 days prior to registration, with the exception of intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection) systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Participants must be >= 18 years of age
* Participants must have Zubrod performance status 0-2
* Participants must have history and physical examination within 28 days prior to registration
* Participants must be surgical candidates as deemed by the local site oncologic surgeon within 28 days prior to registration. This must be clearly documented
* Participants must have a serum creatinine =< the institutional upper limit of normal (IULN) OR measured OR calculated creatinine clearance >= 30 mL/min using the Crockroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* Participants must be deemed cisplatin-ineligible based on greater than or equal to 1 of the following:

  * Zubrod performance status = 2
  * Creatinine clearance (calculated by Crockroft-Gault formula or measured) 30 to < 60 ml/min,
  * Neuropathy > grade 1
  * Hearing loss > grade 1
  * Congestive heart failure > grade 2
* Hemoglobin >= 9.0 g/dL (within 28 days prior to registration)
* Absolute neutrophil count >= 1,500/mcL (within 28 days prior to registration)
* Platelets >= 100,000/mcL (within 28 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to registration)
* Aspartate aminotransferase (AST) =< 2.5 x institutional ULN (within 28 days prior to registration)
* Alanine aminotransferase (ALT) =< 2.5 x institutional ULN (within 28 days prior to registration)
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification and be class 2B or better
* Participants with known human immunodeficiency virus (HIV) must be on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to registration

Exclusion Criteria:

* Participant must not have any other prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, prostate cancer Gleason score =< 3+4 in active surveillance, adequately treated stage I or II cancer from which the participant is currently in complete remission, or any other cancer from which the participant has been disease free for two years
* Participants must not be pregnant or nursing due to the risk of harm to a fetus or nursing infant. Women/men of reproductive potential must have a negative serum or urine pregnancy test within 28 days prior to registration and must have agreed to use an effective contraceptive method. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Participants must not have a history of active primary immunodeficiency
* Participants must not have a history of or active autoimmune or inflammatory disorder, with the exception of vitiligo, alopecia, hypothyroidism (stable on hormone replacement), or chronic skin condition that does not require systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (92):
- United States (92):
  - University of Colorado Hospital, Aurora, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Anthony's Health, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Avelumab, Gemcitabine, Carboplatin, Surgery) | Arm B (Surgery)
Started | 3 | 3
Completed | 3 | 0
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1
Not completed — Not protocol specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Avelumab, Gemcitabine, Carboplatin, Surgery) | Arm B (Surgery) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: Years] | 78 [72 to 79] | 75 [75 to 84] | 76.5 [72 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic: Yes | 0 | 0 | 0
  Hispanic: No | 3 | 3 | 6
  White: Yes | 3 | 3 | 6
  White: No | 0 | 0 | 0
Clinical Stage [Count of Participants; unit: Participants]
  cT2N0M0 | 2 | 3 | 5
  cT3-4aN0M0 | 1 | 0 | 1
Performance Status [Count of Participants; unit: Participants] — 0- Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0-1 | 3 | 3 | 6
    2 | 0 | 0 | 0
Creatinine Clearance [Count of Participants; unit: Participants]
  0 to < 60 ml/min | 1 | 1 | 2
  = 60 ml/min | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: Compare pathologic complete response (pCR) between arms. pCR is defined as s absence of all disease in the surgical specimen from radical cystectomy, nephroureterectomy or ureterectomy as determined by the pathologist at the institution. This is determined by a biopsy taken at the time of surgery.
Time Frame: Measured once - at the time of surgery
Population: Study accrued 6 participants and only 3 participants underwent surgery - 1 in the surgery only arm and 2 in the avelumab, gemcitabine, carboplatin, surgery arm. Thus, pathological response data was only available for the 3 participants who received surgery. There is insufficient data for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Avelumab, Gemcitabine, Carboplatin, Surgery) | Arm B (Surgery)
Number analyzed (Participants) | 2 | 1
Participants
  Complete Response (CR) | 1 | 0
  Stable Disease (STA) | 1 | 0
  Incomplete (INC) | 0 | 1

2. Secondary Outcome: Event-free Survival
Description: Compare event-free survival between arms. Event-free survival is defined as the time from randomization to the first EFS event. For those who do not undergo surgery, event time will be assigned to the date of disease assessment that indicated surgery was no longer indicated or physician decision not to conduct the surgery.
Time Frame: From randomization to the first event, assessed up to study closure
Population: Study only accrued 6 participants and only 3 participants received treatment. Due to lack of data, this objective can not be analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Arm A (Avelumab, Gemcitabine, Carboplatin, Surgery) | Arm B (Surgery)
Number analyzed (Participants) | 2 | 1
days | 349 [217 to 481] | 22 [22 to 22]

3. Secondary Outcome: Incidence of Adverse Events
Description: Evaluate toxicities on both arms. Number of participants with Grade 3-5 adverse events that are possibly, probably or definitely related to study drug are reported. Measured using CTCAE v5.0.
Time Frame: treatment start to 90 days post surgery
Population: Study only accrued 6 participants and only 3 participants received treatment. The three participants who received treatment were assessable for AEs
Measure: Number; unit: Participants
Groups:
- Gemcitabine + Carboplatin + Avelumab + Surgery: Participants receive gemcitabine and carboplatin every 3 weeks for up to 4 cycles and avelumab every 2 weeks for up to 6 cycles, followed by radical cystectomy, nephroureterectomy, or ureterectomy
- Surgery Only: Participants receive radical cystectomy, nephroureterectomy, or ureterectomy
Arm/Group | Gemcitabine + Carboplatin + Avelumab + Surgery | Surgery Only
Number analyzed (Participants) | 2 | 1
Participants
  Neutrophil count decreased | 1 | 0
  Platelet count decreased | 1 | 0

4. Secondary Outcome: Overall Survival
Description: To compare overall survival between arms. Overall survival is defined as time from date of registration to date of death due to any cause or patients last known to be alive are censored at their last contact date.
Time Frame: Up to 5 years post-surgery
Population: Study only accrued 6 participants and only 3 participants received treatment. Because of the study's early termination, there was no data collected for this outcome.
Arm/Group | Arm A (Avelumab, Gemcitabine, Carboplatin, Surgery) | Arm B (Surgery)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pathologic Complete Response - After 2 Cycles
Description: Compare pathologic complete response (pCR) between surgery only arm and participants in the avelumab, gemcitabine, carboplatin, surgery arm who received at least two cycles of treatment. pCR is defined as s absence of all disease in the surgical specimen from radical cystectomy, nephroureterectomy or ureterectomy as determined by the pathologist at the institution. This is determined using a biopsy taken at the time of surgery.
  This outcome uses a subset of participants in arm A who completed exactly 2 cycles of neoadjuvant treatment.
Time Frame: Measured once - at the time of surgery
Population: Study accrued 6 participants and only 3 participants underwent surgery - 1 in the surgery only arm and 2 in the avelumab, gemcitabine, carboplatin, surgery arm. Thus, pathological response data was only available for the 3 participants who received surgery. Both participants in the avelumab, gemcitabine, carboplatin, surgery arm completed at least two cycles of treatment. There is insufficient data for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Avelumab, Gemcitabine, Carboplatin, Surgery) | Arm B (Surgery)
Number analyzed (Participants) | 2 | 1
Participants
  Complete Response (CR) | 1 | 0
  Stable Disease (STA) | 1 | 0
  Incomplete (INC) | 0 | 1

ADVERSE EVENTS:
Time Frame: Treatment start to 90 days post surgery
Description: 3 eligible participants who received at least one dose of protocol treatment were evaluable for Adverse Events (AEs): 2 on the Gemcitabine + Carboplatin + Avelumab + Surgery arm and 1 on the Surgery Only arm. Adverse Events (AEs) and Serious Adverse Events (SAEs) are reported by CTCAE Version 5.0.
Groups:
- Gemcitabine + Carboplatin + Avelumab + Surgery: Participants receive gemcitabine and carboplatin every 3 weeks for up to 4 cycles and avelumab every 2 weeks for up to 6 cycles, followed by radical cystectomy, nephroureterectomy, or ureterectomy.
  Of the 3 participants assigned to this arm, 2 were eligible and included in the at-risk for all cause mortality population. The two participants who receive treatment are included in the at risk for adverse events population.
- Surgery Only: Participants receive radical cystectomy, nephroureterectomy, or ureterectomy.
  Of the 3 participants assigned to this arm, all were eligible and included in the at-risk for all cause mortality population. 1 participant on this arm receive protocol treatment and is included in the at risk for adverse events population.
Arm/Group | Gemcitabine + Carboplatin + Avelumab + Surgery | Surgery Only
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Carboplatin + Avelumab + Surgery (N=2) | Surgery Only (N=1)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vascular disorders-Other (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT04871529/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT04871529/ICF_001.pdf